CLINICAL TRIAL: NCT02500940
Title: Comparison the Effects of Different Neoadjuvant Chemotherapy Regimen on Acute Toxicity, Tumor Response, and Survival in Patients With Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF15113A
Record Dates: First submitted 2015-06-22; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil; Radiotherapy; Leucovorin

ARMS (2):
- Control group (Experimental): Neoadjuvant chemotherapy with tri-weekly cisplatin plus fluorouracil × 3 cycles (cisplatin 100 mg/m2, day 1, followed by fluorouracil 1000 mg/m2/d, days 1-4 continuous iv infusion, repeated every 3 weeks) + Intensity-Modulated Radiation Therapy ≧ 70 Gy/35 fractions
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiation therapy
- Test group (Active Comparator): Neoadjuvant chemotherapy with weekly cisplatin, fluorouracil and leucovorin × 10 weeks (cisplatin 60 mg/m2 at days 1, 15, 29, 43, 57; alternatively with fluorouracil 2500 mg/m2 + leucovorin 250 mg/m2 at days 8, 22, 36, 50, 64) + Intensity-Modulated Radiation Therapy ≧ 70 Gy/35 fractions
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiation therapy; Drug: Leucovorin

INTERVENTIONS:
Drug: Cisplatin — Neoadjuvant chemotherapy regimen with cisplatin
  Other Names: CDDP
Drug: Fluorouracil — Neoadjuvant chemotherapy regimen with Fluorouracil
  Other Names: 5-FU
Radiation: Radiation therapy — Intensity-Modulated Radiation Therapy
  Other Names: IMRT
Drug: Leucovorin — Neoadjuvant chemotherapy regimen with Leucovorin
  Other Names: Calcium folinate
  Arms: Test group

SUMMARY:
The purpose of this study is to investigate the impact of different neoadjuvant chemotherapy schedules of cisplatin and 5-FU on acute toxicity, tumor response, and long-term survival in patients with advanced nasopharyngeal carcinoma

DETAILED DESCRIPTION:
Control group: Neoadjuvant chemotherapy with tri-weekly PF × 3 cycles (cisplatin 100 mg/m2, day 1, followed by 5-FU 1000 mg/m2/d, days 1-4 continuous iv infusion, repeated every 3 weeks) + IMRT ≧ 70 Gy/35 fractions

Test group: Neoadjuvant chemotherapy with weekly P-FL × 10 weeks (cisplatin 60 mg/m2 at days 1, 15, 29, 43, 57; alternatively with 5-FU 2500 mg/m2 + Leucovorin 250 mg/m2 at days 8, 22, 36, 50, 64) + IMRT ≧ 70 Gy/35 fractions

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven NPC.
2. 2010 AJCC stage II-IVB.
3. Age ≧ 20 years old.
4. Performance status of ECOG ≦ 2.
5. Adequate liver, renal, and bone marrow functions 5-1 Serum total bilirubin level ≦ 2.5 mg/dl. 5-2 Serum creatinine ≦ 1.6 mg/dl or calculated CCr ≧ 60 cc/min. 5-3 WBC ≧ 3,000/ul 5-4 Platelet count ≧ 100,000/ul
6. Signed informed consent.

Exclusion Criteria:

1. Presence of distant metastasis.
2. Previous radiotherapy or chemotherapy.
3. History of a malignancy except those treated with curative intent for skin cancer (other than melanoma), in situ cervical cancer, ductal carcinoma in situ (DCIS) of the breast.
4. Severe cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the last 12 months; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders.
5. Female patients who are pregnant or lactating.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Tumor response by RECIST version 1.1 | 5 years
  According to RECIST version 1.1
Overall survival | 5 years

SECONDARY OUTCOMES:
Acute toxicity by CTCAE deifnition | 6 months
  According to CTCAE deifnition

CONTACTS AND LOCATIONS:
Overall Officials: Lin Jin-Ching, Ph.D, Study Chair — Taichung Veterans General Hospital
Locations (1):
- Taichung Vaterans General Hospital, Taichung, Taiwan